CLINICAL TRIAL: NCT05421858
Title: An Interventional Efficacy and Safety Phase 3 Double-blind 2-arm Study to Investigate IV Followed by Oral Fosmanogepix Compared With IV Caspofungin Followed by Oral Fluconazole in Adult Participants With Candidemia and/or Invasive Candidiasis
Brief Title: A Phase 3 Efficacy and Safety Study of Fosmanogepix for the Treatment of Adult Participants With Candidemia and/or Invasive Candidiasis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMGX-CS-301; 2022-500455-23-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT06433128 (Available)
Record Dates: First submitted 2022-06-07; First posted 2022-06-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Candidemia; Candidiasis, Invasive
Keywords: Fungal infection; Candida; Anti-fungal; Yeast
MeSH Terms: conditions — Candidemia; Candidiasis, Invasive; Mycoses; Torulopsis | interventions — Caspofungin; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fosmanogepix IV/oral (Experimental): Fosmanogepix will be administered as an Intravenous (IV) infusion given directly into a vein. There is an option to switch from the IV infusion to the oral form of fosmanogepix which is taken by mouth.
  Matching placebos for caspofungin and fluconazole will also be administered (a placebo does not have any medicine in it but looks just like the caspofungin and fluconazole).
  Interventions: Drug: Fosmanogepix; Drug: Placebo
- Caspofungin IV/ Fluconazole oral (Active Comparator): Caspofungin will be administered as an intravenous (IV) infusion given directly into a vein. There is an option to switch from the IV infusion to oral fluconazole which is taken by mouth.
  Matching placebos for fosmanogepix will also be administered (a placebo does not have any medicine in it but looks just like the medicine fosmanogepix being studied).
  Interventions: Drug: Caspofungin; Drug: Fluconazole; Drug: Placebo

INTERVENTIONS:
Drug: Fosmanogepix — IV infusion
  Arms: Fosmanogepix IV/oral
Drug: Fosmanogepix — Oral tablet
  Arms: Fosmanogepix IV/oral
Drug: Caspofungin — IV infusion
  Arms: Caspofungin IV/ Fluconazole oral
Drug: Fluconazole — Fluconazole oral capsule
  Arms: Caspofungin IV/ Fluconazole oral
Drug: Placebo — Matching placebo for caspofungin (IV infusion)
  Arms: Fosmanogepix IV/oral
Drug: Placebo — Matching placebo for fluconazole (oral capsule)
  Arms: Fosmanogepix IV/oral
Drug: Placebo — Matching placebo for fosmanogepix (IV infusion)
  Arms: Caspofungin IV/ Fluconazole oral
Drug: Placebo — Matching placebo for fosmanogepix (oral tablet)
  Arms: Caspofungin IV/ Fluconazole oral

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called Fosmanogepix) for the potential treatment of candidemia and/or invasive candidiasis, a life-threatening fungal infection caused by several species of yeast called Candida.

The study is seeking patients who have a diagnosis of candidemia and/or invasive candidiasis.

Two-thirds of all patients will receive the study medication fosmanogepix Intravenous (IV) infusion followed by optional fosmanogepix tablets. One-third of all patients will receive a standard of care regimen of caspofungin Intravenous (IV) infusion followed by optional fluconazole capsules.

Fosmanogepix or caspofungin will first be given as an Intravenous (IV) infusion directly into a vein in the arm each day at the study clinic. Fosmanogepix tablets or fluconazole capsules will be taken orally by mouth daily either at the study clinic, or at home if patients are well enough to be discharged from the hospital.

The treatment effect in patients receiving fosmanogepix to those receiving caspofungin/ fluconazole will be compared. The primary aim is to show that fosmanogepix is not inferior (not worse) to caspofungin/ fluconazole with a noninferiority margin of 15%.

The duration of study treatment and number of study visits will vary depending on how long the patient will be treated for the infection. Treatment will continue for a maximum of 6 weeks depending on when the infection is cleared and whether other symptoms related to the infection have improved. There will also be a follow-up visit 6 weeks after the study treatment was stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years (or the minimum country-specific age of consent if > 18) at Screening who have provided signed informed consent indicating that they understand the purpose of, and procedures required for, the study, and are willing to participate in the study. If the patient is unable to consent for himself/herself, a legally authorized representative must provide informed consent on his/her behalf.
2. Diagnosis of candidemia and/or invasive candidiasis based on a blood or non-blood specimen obtained within ≤ 96 hours (4 days) before randomization, and on clinical criteria judged attributable to candidemia/invasive candidiasis occurring at any time from ≤ 12 hours prior to the qualifying positive index culture being taken through to randomization.
3. Patient's condition allows for appropriate infection source control measures, including removal of pre-existing intravascular catheters and devices, if necessary.

Exclusion Criteria:

1. Existing infection

   1. Infection known to be due to Candida krusei, in blood or any other normally sterile site.
   2. Inappropriate fungal infection source control.
   3. Diagnosis of certain deep-seated Candida infections.
2. Life expectancy of < 72 hours in the opinion of the investigator.
3. Requirement, or expected requirement, for hemodialysis, peritoneal dialysis, or hemofiltration.
4. Ongoing neurological disorders, including specified conditions presenting with a CTCAE Grade ≥ 2 (neurological symptoms that are considered to be a consequence of the current episode of candidemia / invasive candidiasis are not exclusionary).
5. Patients with known human immunodeficiency virus infection, who have CD4+ count < 200/mm3 or viral load > 400 copies/mL), or who have had an active opportunistic infection within 6 months prior to Screening.
6. Other medical or psychiatric condition or laboratory abnormality that may increase the risk of study participation or make the patient inappropriate for the study.
7. Current use of any prohibited concomitant medications or those unwilling/unable to use a permitted concomitant medication.
8. Received > 2 days (> 48 hours) equivalent of prior systemic antifungal treatment at approved doses and frequency to treat the current episode of candidemia and/or invasive candidiasis (e.g., > 2 doses of a once daily antifungal agent or > 4 doses of a twice daily antifungal agent), within the 96 hours prior to randomization (except for non-susceptible Candida spp. and for patients who develop candidemia or invasive candidiasis while on prophylaxis with an azole or amphotericin B).
9. Previous administration with an investigational drug or investigational vaccine within 30 days or 5 half-lives preceding the first dose of study drug used in this study (whichever is longer).
10. Prior participation in this or any previous study of fosmanogepix.
11. Moderate or severe hepatic impairment, known active viral hepatitis B or C, ALT or AST ≥ 5 × ULN or total bilirubin > 3 × ULN unless this is due to isolated hyperbilirubinemia or documented Gilbert's syndrome.
12. Female patient is pregnant or lactating.
13. Known hypersensitivity to fosmanogepix, manogepix, caspofungin, any echinocandin, fluconazole or to any of their excipients.
14. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and Sponsor and Sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients alive at Day 30 | Day 30
Proportion of patients with an overall response of treatment success at end of study treatment (EOST) | EOST (up to Day 42)

SECONDARY OUTCOMES:
Proportion of patients with an overall response of treatment success at Day 7 | Day 7
Proportion of patients with an overall response of treatment success at Day 14 | Day 14
Proportion of patients with an overall response of treatment success at end of IV treatment (EOIV) | up to Day 42
Proportion of patients with an overall response of treatment success (sustained) at follow-up 6 weeks after EOST | approximately up to 12,5 weeks
Proportion of patients with clinical response of success at Day 7, 14, EOIV, EOST, Follow-up 6- weeks after EOST | Day 14, EOIV (up to Day 42), EOST (up to Day 42), Follow-up 6-weeks after EOST]
Proportion of patients with mycological response of eradication or presumed eradication at Day 7, 14, EOIV, EOST, Follow-up 6-weeks after EOST | Day 14, EOIV (up to Day 42), EOST (up to Day 42), Follow-up 6-weeks after EOST
Time to first negative blood culture in patients on fosmanogepix compared to caspofungin/fluconazole | Baseline up to follow-up 6-weeks after EOST (approximately up to 12,5 weeks)
Incidence of treatment-emergent adverse event (TEAEs), serious adverse events (SAEs), treatment-related adverse events (AEs), adverse events of special interest (AESI)and AEs leading to discontinuation | Screening up to follow-up 6-weeks after EOST (approximately up to 12,5 weeks)
Number of patients with clinically significant laboratory abnormalities | Baseline up to follow-up 6-weeks after EOST (approximately up to 12,5 weeks)
Number of patients with abnormal neurological examination findings | Baseline up to follow-up 6-weeks after EOST (approximately up to 12,5 weeks)
Assessment of 12-lead electrocardiogram (ECGs) | Baseline up to follow-up 6-weeks after EOST (approximately up to 12,5 weeks)
Plasma concentrations versus time of fosmanogepix (prodrug) and manogepix (active moiety) | Day 3: 0, 3, 6, 9 and 24 hours post-dose; Day 7, 14, 21, 28, 35; EOST: 72 and 192 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Häckl, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (110):
- United States (15):
  - University of Alabama at Birmingham School of Medicine, Department of Medicine, Birmingham, Alabama
  - UC Davis Medical Center, Sacramento, California
  - Emory University Hospital - Clifton Road, Atlanta, Georgia
  - Indiana University Methodist Hospital, Indianapolis, Indiana
  - University of Kentucky College of Medicine, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Health System (UMHS) - A. Alfred Taubman Health Care Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Department of Medicine, Division of Infectious Diseases, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, Infectious Diseases Clinical Research Unit, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Houston Methodist Hospital - Texas Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Carilion Clinic, Roanoke, Virginia
- Argentina (6):
  - Central Hospital de San Isidro Melchor Posse, Buenos Aires
  - Buenos Aires Italian Hospital, Department of Infectious Diseases, Buenos Aires
  - Cordoba Private University Hospital, Department of Infectious Diseases, Córdoba
  - Italian Hospital of La Plata, Department of Infectious Diseases, La Plata
  - Central Hospital Mendoza, Mendoza
  - British Sanatorium SA, Rosario
- Australia (6):
  - Westmead Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Center, State, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Monash Medical Center Clayton, Clayton
- Austria (4):
  - University Hospital Graz, Department of Internal Medicine, Graz
  - Kepler University Hospital GmbH, Department of Pulmonology, Clinical Department of Infectious Diseases, Linz
  - Medical University Vienna, Vienna
  - Hospital Favoriten, Department of Internal Medicine IV - Infectious Diseases and Tropical Medicine, Vienna
- Belgium (7):
  - General Hospital Saint-Jan, Bruges
  - University Hospital Brussels, Brussels
  - Saint Luc University Hospital, Department of Internal Medicine, Brussels
  - Erasme Hospital, Department of Infectious and Tropical Diseases, Brussels
  - Jessa Hospital, Hasselt
  - University Hospitals Leuven, Campus Gasthuisberg, Department of Infectious Diseases, Leuven
  - UCL Mont-Godinne University Hospitals, Yvoir
- Brazil (4):
  - Hospital Our Lady of Grace, Curitiba, Paraná
  - Porto Alegre Clinical Hospital (HCPA), Infectious Diseases / Internal Medicine, Porto Alegre, Rio Grande do Sul
  - Pontifical University Of Rio Grande Do Sul (PUCRS) - St. Luke Hospital, Porto Alegre, Rio Grande do Sul
  - Santa Marcelina Hospital, São Paulo
- Bulgaria (3):
  - Eurohospital University Hospital, Plovdiv
  - University Medical Center "N. I. Pirogov", Burns and Plastic Surgery Clinic, Sofia
  - University Medical Center "N. I. Pirogov", Clinic of Purulent-Septic Surgery, Sofia
- Somer Clinic, Rionegro, Colombia
- France (6):
  - Amiens Picardie University Hospital - South, Intensive Care Unit (ICU), Amiens
  - Victor Dupouy Hospital Center Argenteuil, Intensive Care Unit, Argenteuil
  - Marseille Nord University Hospitals - AP-HM, Medical Intensive Care Unit, Acute Respiratory Distress and Severe Infections, Marseille
  - Nantes University Hospital Center - Hotel Dieu Hospital, Department of Infectious and Tropical Diseases, Nantes
  - Rennes University Hospital Center - Hospital Pontchaillou, Rennes
  - Tours Regional University Hospital Center, Tours
- Germany (6):
  - University Hospital Ulm, Comprehensive Infectious Diseases Center Ulm (CIDCU), Ulm, Baden-Wurttemberg
  - University Hospital Regensburg, Regensburg, Bavaria
  - Frankfurt University Clinic, Frankfurt am Main, Hesse
  - University Hospital Giessen and Marburg GmbH, Giessen, Hesse
  - University Hospital Cologne, Department of Internal Medicine I, Clinical Study Centre II for Infectious Diseases, Cologne, North Rhine-Westphalia
  - University Hospital Heidelberg, Clinic for Anesthesiology, Heidelberg
- Greece (5):
  - "LAIKO" General Hospital, Athens
  - "Sotiria" Chest Diseases Hospital of Athens, Athens
  - General Hospital of Athens "Evangelismos", 5th Department of Internal Medicine and Infectious Diseases Unit, Athens
  - Tzaneio General Hospital, Piraeus
  - General Hospital of Thessaloniki "Ippokratio", Thessaloniki
- Israel (5):
  - Rambam Health Care Campus, Institute of Infectious Diseases, Haifa
  - Edith Wolfson Medical Center, Department of Infectious Diseases, Holon
  - Chaim Sheba Medical Center, Department of Infectious Diseases, Ramat Gan
  - The Tel Aviv Sourasky Medical Center, Infectious Diseases Unit, Tel Aviv
  - Shamir Medical Center, Department of Infectious Diseases, Ẕerifin
- Italy (10):
  - Hospital "S. Croce e Carle", Cuneo
  - IRCCS Policlinic Hospital San Martino, Genoa
  - Maggiore Polyclinic Hospital, Foundation IRCCS Ca' Granda, Milan
  - Hospital San Raffaele, IRCCS, Milan
  - Big Metropolitan Hospital Niguarda Regional Health Authority, Milan
  - University Polyclinic Hospital of Modena, Modena
  - Polyclinic San Matteo, IRCCS, Pavia
  - University Hospital of Pisa, Pisa
  - AOU Senese, Siena
  - Giuliano Isontina University Health Authority, Trieste
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Africa (5):
  - Helen Joseph Hospital, Johannesburg
  - Milpark Hospital, Johannesburg
  - Ryexo Clinical Research, Pretoria
  - University of Pretoria / Steve Biko Academic Hospital, Pretoria
  - Practice of R Moodley and MI Sarvan - Umhlanga, Umhlanga
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (7):
  - University Hospital Virgen Macarena, Seville, Andalusia
  - University Hospital Nuestra Senora de Valme, Seville, Andalusia
  - Hospital del Mar, Department of Infectious Diseases, Barcelona, Catalonia
  - University Hospital Vall d'Hebron, Intensive Care Unit (ICU), Barcelona, Catalonia
  - Hospital Clinic of Barcelona, Department of Infectious Diseases, Barcelona, Catalonia
  - University Hospital Ramon y Cajal, Department of Infectious Diseases, Madrid, Madrid
  - University Hospital Cruces, Barakaldo
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- Thailand (5):
  - Vajira Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Khon Kaen

IPD SHARING:
Plan to Share IPD: No